CLINICAL TRIAL: NCT00819364
Title: Early Intervention Program for Children With Autism (BCRI Model)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-sen University (Other)
Responsible Party: The Third Affliated Hospital of Sun Yat-sen University, The Third Affliated Hospital of Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007024
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: Autism; early intervention; BCRI model
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants with autism will receive BCRI intervention program.
  Interventions: Behavioral: BCRI intervention program
- 2 (Active Comparator): Participants with autism will receive standard care available in the community.
  Interventions: Behavioral: Standard community care

INTERVENTIONS:
Behavioral: BCRI intervention program — Phase 1: The parents will receive a two-day lecture about autism to get the basic knowledge about autism intervention.
  Phase 2: BCRI model intervention.Parents and children will take part in a 24-halfday workshop to learn practical teaching skills in BCRI model. Then Home-based intervention using BCRI model for 11 months. At least 28 hours of BCRI intervention per week is acquired. Doctors or therapists will meet the parents and children once per month, each for 30 minutes, totally 10 times, to monitor and give advice on the interventions.
  Arms: 1
Behavioral: Standard community care — Phase 1: the parents will receive a two-day lecture about autism to get the basic knowledge about autism intervention.
  Phase 2:Any treatment and interventions available chosen by families for children with autism and ASD, for at least one and a half years.
  Phase 3:One and a half years after enrollment, parents and children will be free to take part in the BCRI model intervention which is the same as Phase 2 for experimental group lasting for one year.
  Arms: 2

SUMMARY:
This is a randomized controlled study to determine whether the BCRI (Behavior-Cognition-Relationship Intervention) model is effective for the autistic children. BCRI model is a eclectic method using behavior modification, structure teaching, relationship-focus approaches according to the symptom severity and main problems at any stage of training for the autistic children. The BCRI Model emphasis the importance that parents understand the principle of training and education and can use them skillfully, appropriately and persistently.

DETAILED DESCRIPTION:
In recent years, autism has been found that the outcomes can be much better after early training interventions. The training programs are often categorized as behavior analytic, cognitive or structured teaching, developmental or relationship-focused and so on. Although the approaches focus on different aspect of rehabilitation, they also overlap, playing complementation roles for one another. From our clinical experiences, we find that different children, in their different stages, with different problems, will need different approaches. For example, at early stage behavior modulation method is useful to regulate the child's behaviors. When the child is able to cooperate with adults, structure teaching helps him/her improve cognitive ability. Relationship-focused methods may help the child on social interaction. BCRI model, a comprehensive model, is based on the three kinds of approaches above.

All the autistic children will receive examinations before assignment, including history and symptoms collection, diagnostic interview, evaluation(using PEP-3 for autistic children to evaluate intelligence level). DQ is calculated through PEP-3 assessment. (DQ, development quotient, equals to development age in month over chronological age in month). Children will be randomly assigned to one of two interventions arms: BCRI intervention program or standard community care.

BCRI intervention program aims to teach the parents to master how to apply correct approaches and strategies and hold the training both at home and/or in training institutes. During the program, doctors deliver the knowledge and skills to the parents, set a complete schedule for the intervention, assess the progress and development for the children and communicate with the parents about any problems and frustration. Parents play an important and direct role in the training and educating procedure. The contrast group receives standard community intervention.

ELIGIBILITY:
Inclusion Criteria for Autistic Participants:

* younger than 30-month old
* must be diagnosed as Autism Spectrum Disorder（autism, PDD-NOS, Asperger's disorder）according to the diagnostic criteria in DSM-IV, or showing symptoms that child may be developing autism.
* Within 2 hour drive of the third affiliated hospital of SUMS.
* Willing to participate in either of 2 randomly assigned treatment groups and carry out the intervention as advices. Attendance at all activities and sessions.
* Both of the parents at least get a high school degree.

Exclusion Criteria:

* Rett syndrome.
* mental retardation associated with brain injury, fragile X syndrome, tuberous sclerosis, phenyl ketonuria, phenyl ketonuria, Angelman syndrome、Prader-Willi syndrome and autism accompanied with sensory or motor impairments.

Max Age: 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2009-08; Primary Completion 2013-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Psychoeducational Profile-3rd Edition(PEP-3) | Measured before and after treatment and at 2-year follow-up

SECONDARY OUTCOMES:
SRS(social response scale) scores and/or C-WYCSI scores at 2-year follow-up. SRS(social response scale) scores and/or C-WYSC scores at 5-year follow-up. | Measured at 2-year and 5-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Zou Xiaobing, M.D., Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University